CLINICAL TRIAL: NCT00261534
Title: Outcomes Research on the Course of Cancer Related Fatigue Throughout Five Chemotherapy Treatments
Brief Title: Cancer Related Fatigue in Patients Receiving Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical Center Alkmaar (Other)
Other Study IDs: M05-057
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Cancer; Fatigue
Keywords: Chemotherapy
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examine the degree of fatigue in patients receiving chemotherapy. Special interest goes out to the course of fatigue throughout five treatments and the actions taken by patients to reduce this fatigue.The correlation between fatigue and haemoglobin will also be subject of study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer requiring chemotherapy treatment

Exclusion Criteria:

* Pregnancy
* Psychological illness
* Life expectancy less than three months
* Lack of basic proficiency in Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: D. Hilarius, MSc, Study Director — Medical Centre Alkmaar, Hospital Pharmacy
Locations (1):
- Medical Centre Alkmaar, Alkmaar, North Holland, Netherlands